CLINICAL TRIAL: NCT07130578
Title: Truce-LB00:The Guiding Value of Liquid Biopsy Based on Urinary Tumor DNA/RNA in the Second Transurethral Resection of High-risk Non-muscle Invasive Bladder Cancer: An Open-Label, Observational, Single-Center Clinical Study
Brief Title: The Guiding Value of Liquid Biopsy Based on Urinary Tumor DNA/RNA in the Second Transurethral Resection of High-risk Non-muscle Invasive Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Truce-LB00
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer; Liquid Biopsy
Keywords: Bladder Cancer; Liquid Biopsy; NMIBC; re-TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The genes of tumor exfoliated cells in urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All enrolled patients will undergo urine tumor DNA (utDNA) and urine tumor RNA (utRNA) testing between 2-6 weeks after the initial transurethral resection of bladder tumor (TURBT) and prior to the second TURBT (re-TURBT). The re-TURBT procedure will include deep resection at the site of the original tumor base, complete resection of tumor margins and any suspicious areas, as well as random bladder biopsies as indicated. The results of utDNA/utRNA testing will be compared with pathological findings from the re-TURBT specimens to evaluate the diagnostic value of molecular urine testing in detecting residual disease.
  Interventions: Diagnostic Test: urine tumor DNA/RNA testing

INTERVENTIONS:
Diagnostic Test: urine tumor DNA/RNA testing — The test analyzes DNA and RNA fragments shed by urothelial carcinoma cells into urine, detecting tumor-specific genetic and epigenetic alterations.

SUMMARY:
High-risk non-muscle-invasive bladder cancer (NMIBC) carries a substantial risk of residual disease after initial transurethral resection of bladder tumor (TURBT). Current guidelines recommend a second TURBT (re-TURBT) within 2-6 weeks for patients with stage T1 disease to remove residual tumor, confirm staging, and obtain additional pathological information. However, the actual survival benefit of routine re-TURBT for all high-risk patients remains debated, and the procedure may pose surgical risks, increase healthcare costs, and impact patient quality of life.

Urine tumor DNA (utDNA) and urine tumor RNA (utRNA) are molecular biomarkers detectable through non-invasive "liquid biopsy" methods. In urothelial carcinoma, tumor-derived nucleic acids can be shed into urine, where they can be detected with high sensitivity and specificity. These biomarkers may help identify patients most likely to harbor residual disease after initial TURBT, and thus most likely to benefit from re-TURBT.

This prospective, open-label, observational, single-center study aims to evaluate the clinical value of utDNA/utRNA testing in guiding re-TURBT for patients with high-risk NMIBC. The study will assess whether molecular urine testing can improve patient selection for re-TURBT, potentially reducing unnecessary procedures while maintaining oncological safety.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the study:

1. Male or female, aged 18 years or older.
2. Histologically confirmed non-muscle-invasive bladder tumor, with no evidence of muscle-invasive bladder cancer or metastatic disease.
3. Histologically confirmed urothelial carcinoma of the bladder or bladder tumor with urothelial carcinoma as the predominant component (>50%).
4. At least one of the following conditions:

   1. Incomplete initial transurethral resection of bladder tumor (TURBT) or suspected incomplete resection.
   2. Absence of detrusor muscle in the initial TURBT pathological specimen (except for low-grade Ta stage tumors or carcinoma in situ [CIS]).
   3. T1 stage tumor.
5. Willingness to provide a 50 mL urine sample between 2-6 weeks after the initial TURBT and prior to re-TURBT.
6. Willingness to provide tumor tissue samples for pathological examination.
7. Willingness to undergo genetic testing required for the trial.
8. Voluntarily agrees to participate in the study, has signed informed consent, demonstrates good compliance, and is willing to complete study follow-up.

Exclusion Criteria:

1. Contraindications to transurethral resection of bladder tumor (TURBT).
2. Concurrent malignancy of the upper urinary tract (ureter or renal pelvis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with histologically confirmed high-risk non-muscle-invasive bladder cancer (NMIBC) who have undergone initial transurethral resection of bladder tumor (TURBT) and are scheduled for second TURBT. Eligible tumors are urothelial carcinoma or bladder tumors with urothelial carcinoma as the predominant component (>50%), with no evidence of muscle-invasive or metastatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Concordance analysis of urine tumor DNA/RNA testing results with results of secondary TURBT histopathology | Through study completion, an average of 6 months
  Through Concordance analysis of urine tumor DNA/RNA testing results with gold standard results of secondary TURBT histopathology, the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Tianjin Medical University, Tianjin, China

IPD SHARING:
Plan to Share IPD: No